CLINICAL TRIAL: NCT04111588
Title: Diagnostic Assessment of Amino Acid PET/MRI in the Evaluation of Glioma and Brain Metastases
Status: Recruiting | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); University of Bergen (Other); Haukeland University Hospital (Other); University of Tromso (Other); University Hospital of North Norway (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/2243
Record Dates: First submitted 2019-09-28; First posted 2019-10-01 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-05

CONDITIONS: Brain Neoplasms
Keywords: Diagnosis; Magnetic Resonance Imaging; Positron-Emission Tomography; PET-tracer
MeSH Terms: conditions — Brain Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Glioma: 20 low-grade (LGG) and 40 high-grade glioma (HGG) patients will be included from the Department of Neurosurgery at St. Olavs Hospital and the Department of Neurosurgery at the University hospital of North Norway and examined with 18F-FACBC PET/MRI at baseline and 4-6 months after surgery. Furthermore, 10 of the LGG patients and 10 of the HGG patients will be examined with an additional 18F-FET PET/MRI at baseline for comparison with 18F-FACBC.
  30 recurrent HGG patients will be recruited from the Department of Neurosurgery and the Department of Oncology at the Haukeland University Hospital. These patients will be examined with 11C-MET PET/MRI at treatment/baseline and 1 month after radiosurgery.
  Interventions: Other: Diagnostic Amino acid PET/MRI examination
- Brain Metastases: Patients with brain metastases (18F-FACBC: n=20, 18F-FET: n=20 and 11C-MET: n=30) will be included from the Department of Neurosurgery at St. Olavs Hospital, the Department of Neurosurgery at Haukeland University Hospital and the Department of Neurosurgery at the University hospital of North Norway, and examined with amino acid PET/MRI at baseline, 1 month after surgery/stereotactic radiosurgery (St. Olavs Hospital/UNN: Linac, Haukeland University Hospital: Gamma Knife® radiosurgery) and at suspicion of recurrence.
  Interventions: Other: Diagnostic Amino acid PET/MRI examination

INTERVENTIONS:
Other: Diagnostic Amino acid PET/MRI examination — Diagnostic Amino acid PET/MRI examination

SUMMARY:
MRI is used in clinical routine for diagnosing brain tumors, but has limitations in identifying tumor grade, true tumor extension and differentiate viable tumor tissue from treatment induced changes and recurrences.

Amino acid PET has demonstrated a great potential for defining true tumor volume, differentiate viable tumor tissue from postoperative changes or radiation necrosis, selection of biopsy site, non-invasive grading of gliomas and for treatment planning and therapy response assessment. By combining PET with MRI, the diagnostic accuracy can improve significantly for these patients. More research is however needed to compare the most promising amino acid PET tracers in patients with glioma, but also to assess the diagnostic value of amino acid PET in patients with different brain metastases, where the knowledge concerning the uptake characteristics is limited.

Three of the most promising amino acid tracers ([11C]-methyl-methionine (11C-MET), [18F] fluoro-ethyl-tyrosin (18F-FET) and anti-1-amino-3-[18F]fluorocyclobutane-1-carboxylic acid (18F-FACBC)) will be evaluated in 3 substudies in this project; WP1 Aminoacid PET/MRI in low and high grade glioma; WP2 Role of 11C-MET in high-grade glioma Gamma Knife® radiosurgery; and WP3 Amino acid PET in brain metastasis.

The main aim of the study is to improve diagnostic accuracy, histopathological tissue sampling, delineation of tumor extent and therapy response assessment in gliomas and brain metastases with amino acid PET/MRI.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria Glioma (LGG, HGG and recurrent HGG):

  * Planned treatment for WHO grade II-IV diffuse glioma
  * Adult patients (>18 years)
  * Planned tissue sampling for histopathological diagnosis.
  * KPS >60 (able to care for self)

Inclusion criteria Brain Metastasis:

* Indication of surgery or stereotactic radiosurgery for 1-4 brain metastases
* Planned surgery: Suspicion of brain metastasis or known diagnosis
* Stereotactic surgery: Known primary cancer
* Adult patients (>18 years)
* Estimated survival at least 3 months after inclusion

Exclusion Criteria:

* Exclusion criteria (Glioma and Brain Metastasis):

  * Pacemakers or defibrillators not compatible with 3T MRI
  * No ability to obtain informed consent (e.g. due to severe dysphasia or cognitive deficits).
  * Pregnancy (pregnancy test for all women in fertile age when doubt about possible pregnancy exist)
  * Breastfeeding
  * Weight > 120 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * 20 low-grade glioma (LGG) patients
  * 40 high-grade glioma (HGG)
  * 30 recurrent HGG patients
  * 70 Patients with brain metastases
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2019-11-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy in detecting brain tumor tissue at baseline | Baseline
  Diagnostic accuracy, sensitivity, specificity, positive-and negative predictive values of PET, contrast-enhanced MRI (MRICE) and combined PET/MRI will be calculated by comparing images to histopathological results for the large non-localized biopsies as well as to the image-localized biopsies taken prior to resection.

SECONDARY OUTCOMES:
Diagnostic accuracy using dynamic PET | Baseline
  Dynamic PET will be compared for differentiation between low-grade and high-grade tumors and to study the relationship between the time-activity-curve pattern and histology type.
Differentiation between recurrence and treatment related changes using PET/MRI | 4-6 months
  18F-FACBC uptake (at follow-up), in terms of SUV, TBR, and TAC will be compared to MRI and baseline-PET to evaluate if PET can detect recurrent disease prior to MRI, or if PET can define early treatment response better than MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Live Eikenes, Phd, Principal Investigator — Norwegian University of Science and Technology; Øystein Risa, Study Director — Norwegian University for Science and Technology
Locations (3):
- Norway (3):
  - Haukeland universitetssykehus, Bergen
  - Universitetssykehus Nord Norge, Tromsø
  - St Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karlberg A, Pedersen LK, Vindstad BE, Skjulsvik AJ, Johansen H, Solheim O, Skogen K, Kvistad KA, Bogsrud TV, Myrmel KS, Giskeodegard GF, Ingebrigtsen T, Berntsen EM, Eikenes L. Diagnostic accuracy of anti-3-[18F]-FACBC PET/MRI in gliomas. Eur J Nucl Med Mol Imaging. 2024 Jan;51(2):496-509. doi: 10.1007/s00259-023-06437-4. Epub 2023 Sep 30. PMID 37776502
- [Derived] Kotecha R, Aboian M, Nabavizadeh SA, Parent EE, Trifiletti DM, Chao ST. Letter regarding "Contribution of PET imaging to radiotherapy planning and monitoring in glioma patients-a report of the PET/RANO group": 18F-fluciclovine and target volume delineation. Neuro Oncol. 2021 Aug 2;23(8):1408-1409. doi: 10.1093/neuonc/noab097. No abstract available. PMID 34081125